CLINICAL TRIAL: NCT05846386
Title: Effects of Early Resistance Training on Functional Capacity and Electrocardiographic Changes Post Valve Replacement Surgery
Brief Title: Early Resistance Training Post Valve Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: RMIT University, Melbourne, Australia (Unknown); Federation University Australia (Other)
Responsible Party: Principal Investigator, Hady Atef Labib, Lecturer of physiotherapy for cardiovascular/respiratory disorders, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: post valve replacement
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Valve Disease, Heart
Keywords: post valve replacement; resistance exercise; aerobic exercise
MeSH Terms: conditions — Heart Valve Diseases | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic and resistance training (Experimental): aerobic exercises (intervention) on arm ergometer and resistance training using weights for post valve replacement surgery patients for 4 weeks, 3 times/week for the duration of 45-70 min/ session.
  Interventions: Behavioral: Resistance training; Behavioral: Aerobic training
- Aerobic training (Active Comparator): aerobic exercises (intervention) on arm ergometer for post valve replacement surgery patients for 4 weeks, 3 times/week for the duration of 30-55 min/ session.
  Interventions: Behavioral: Aerobic training

INTERVENTIONS:
Behavioral: Resistance training — moderate-intensity resistance training: three sessions per week for one month. Participants had been instructed to perform exercises at a 4:2:4 tempo; that is, four sets of concentric contraction, two sets of isometric hold, and four sets of eccentric contraction. Participants had been instructed to complete a single set until volitional fatigue or been instructed to stop by the physiotherapist when the technique falters
  Arms: Aerobic and resistance training
Behavioral: Aerobic training — The exercise program consisted of ten minutes warm-up, 45 minutes of moderate aerobic exercises "upper extremity aerobic bulk muscles training and arm ergometer" and cool-down in five minutes, respectively. That was done as 3 sessions/week for 4 weeks.

SUMMARY:
Background: Recent recommendations from the European Society of Cardiology (ESC) are multidisciplinary cardiac rehabilitation including therapeutic exercises for patients after heart valve surgery unless there is insufficient evidence to decide whether therapeutic exercise cardiac training should be provided for such patients. As well, resistance training is an extremely safe systemic physical activity, and it has no contraindications if well-oriented, in addition to being the fastest-growing physical activity in the world in several practitioner settings.

Purpose: This study was conducted to investigate the effect of early resistance training on the fitness level (vo2 max) and (PR interval) of patients post-valve replacement surgery.

DETAILED DESCRIPTION:
Method: Forty males post-valve replacement surgery participants' age ranged from 20 to 30 years old and were selected randomly from National Heart Institute (Imbaba), this study was conducted in the period between April and November 2022, and those participants were allocated randomly into two equal groups twenty in each group. Group A received aerobic and resistance training three sessions per week for one-month, and group B received aerobic training three sessions per week for one month. All demographic data was recorded and an ECG device was used to record HR and R-P Intervals, Six-Minute Walk Test (6MWT) was used to assess of cardiorespiratory fitness for all participants in both groups (A&B)

ELIGIBILITY:
Inclusion Criteria:

1. Participants' age ranged from 20 to 30 years old,
2. Participants medically stable to do early resistance exercise in the first week after the operation.
3. Each participant had undergone valve replacement surgeries only,
4. Participants be able to do early resistance exercises in the first week after the operation.

Exclusion Criteria:

* The study excluded the participant if has one or more of the following criteria:

  * sternal infection and delay sternal healing.
  * Patient with a musculoskeletal condition limiting the ability to exercise or a geographical residence and/or lack of access to transportation, thus preventing exercise session attendance.
  * The patient has an LV thrombus diagnosed by echocardiography, left ventriculogram, or other imaging.
  * The patient is known to have unprotected left main coronary artery disease (CAD) greater than 50%.
  * Patients have poor cognitive capabilities or poor mentality.
  * Patient who had valve and CABG surgery.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
six minute walking distance (in meters) | 4 weeks
  represent aerobic capacity (distance walked in 6 min)
P-R interval (in milliseconds) | 4 weeks
  represent a mortality index (the time from the beginning of atrial depolarization to the onset of ventricular depolarization) on the electrocardiograph

CONTACTS AND LOCATIONS:
Overall Officials: Hady Atef, Ph.D., Principal Investigator — Cairo University
Locations (1):
- National heart institute, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After approval can be shared
Supporting Information: Study Protocol
Time Frame: after 1 month for 12 months
Access Criteria: will upload it to the journal of publication